CLINICAL TRIAL: NCT04937777
Title: A Retrospective Observational Multicenter Study on the Management and Outcome of Patients With Systemic AL Amyloidosis in Europe
Brief Title: A Study on the Management and Outcome of Patients With Systemic AL Amyloidosis in Europe
Status: Completed | Type: Observational
Sponsor: European Myeloma Network B.V. (Network)
Responsible Party: Sponsor
Other Study IDs: EMN23
Record Dates: First submitted 2021-04-06; First posted 2021-06-24 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group pre-2010: Patients who initiated first-line treatment between 2004 and 2010 (pre-2010).
- Group post-2010: Patients who initiated first-line treatment between 2011 and 2018 (post-2010).

SUMMARY:
This is a retrospective, observational, multicenter study to collect Real-World Evidence (RWE) data on systemic AL-AMY patients in Europe. Data from paper/electronic medical records and/or electronic databases from key reference centers in Europe will be used. Data will either be entered by the site staff in the electronic Case Report Form (eCRF) or, where feasible, transferred directly, always in accordance to local regulations.

DETAILED DESCRIPTION:
The lack of regulatory approved treatment options for AL amyloidosis (AL-AMY) justifies the need to understand the current treatment practice and outcomes of this disease. There is a need for objective Real-World Evidence (RWE) that reflects how treatments are initiated, combined and sequenced, and how their relative effectiveness and safety profiles emerge outside a clinical trial setting. Therefore, the aim is to generate RWE on systemic AL-AMY patients in Europe, including patient characteristics, resource use, treatments and associated patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Confirmed diagnosis of AL-AMY and symptomatic organ involvement.
* Initiated first line treatment for AL-AMY in the period 2004-2018.
* Patients who have signed a participation agreement/ICF allowing data collection and source data verification in accordance with local requirements.

The inclusion of deceased subjects in the study is permitted under the condition that consent waiver has been granted by the Scientific Committee and/or Administrative Board of the participating sites and/or any applicable regulatory body, as per local regulations, to either implement a hospital informed consent form (ICF) already in place or provide written approval of this study-specific waiver. In the occasion that waiver of consent is not granted deceased subjects will not be enrolled in the study.

Exclusion Criteria:

* Patients under the age of 18 will not be considered eligible for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult (male and female) patients diagnosed with systemic AL-AMY and symptomatic organ involvement who have initiated first line treatment in the period 2004-2018.
  Patients who have received treatment for AL-AMY as part of an interventional Clinical Trial will be identified but will not be included in the analysis due to the controlled environment of a clinical trial (not RWE data).
  Patients with comorbid multiple myeloma will not be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 4481 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Patient and disease characteristics | 2004-2018
  To describe the proportion of patients belonging to different age groups, and the proportion of patients per gender, stage, organ involvement, performance status, and hematologic biomarkers at screening or at baseline; by first-line treatment initiation period (pre-2010 or post-2010) and overall.
Treatment patterns | 2004-2018
  To describe the proportion of patients who had an autologous stem cell transplantation by first-line initiation period (pre-2010 or post-2010) and overall; the proportion of regimen combinations used by line of treatment, and by first-line initiation period; the proportion of patients receiving specific regimen combinations following different first-line regimens, by first-line initiation period and overall.
Response evaluation and efficacy outcomes | 2004-2018
  To describe the treatment effectiveness in terms of hematologic response rates at 3, 6, 12, and 24 months after first-line initiation, by regimen and first-line initiation period (pre-2010 or post-2010); overall survival, progression-free survival, and time on treatment, overall, by first-line treatment and by first-line initiation period.
Healthcare resource utilization: hospitalizations | 2004-2018
  To describe the healthcare resource utilization patterns during the treatment of AL amyloidosis by first-line treatment initiation period (pre-2010 or post-2010) and overall, in terms of hospitalization information (number of hospitalizations, duration per hospitalization); use of concomitant treatment (frequency of regimens used, proportion of patients receiving concomitant treatment); proportion of patients undergoing imaging exams; proportion of patients undergoing cardiac exams; proportion of patients receiving dialysis.
Healthcare resource utilization: concomitant therapy | 2004-2018
  To describe the healthcare resource utilization patterns during the treatment of AL amyloidosis, by first-line treatment initiation period (pre-2010 or post-2010) and overall, in terms of the proportion of patients receiving concomitant therapy.
Healthcare resource utilization: imaging and cardiac assessments | 2004-2018
  To describe the healthcare resource utilization patterns during the treatment of AL amyloidosis, by first-line treatment initiation period (pre-2010 or post-2010) and overall, in terms of the proportion of patients undergoing imaging and cardiac exams.
Healthcare resource utilization: dialysis | 2004-2018
  To describe the healthcare resource utilization patterns during the treatment of AL amyloidosis, by first-line treatment initiation period (pre-2010 or post-2010) and overall, in terms of the proportion of patients receiving dialysis.
Safety management | 2004-2018
  To describe the proportion of patients having serious adverse events or adverse events of special interest, by first-line treatment initiation period (pre-2010 or post-2010) and overall.

CONTACTS AND LOCATIONS:
Locations (13):
- Allgemeines Krankenhaus Der Stadt Wien (General Hopsital), Universitätsklinik Für Innere Medizin I Klinische Abteilung Für Onkologie (Clinic of Internal Medicine I), Medizinische Universität Wien, Vienna, Austria
- University Hospital Ostrava, Clinic of Hematooncology, Ostrava, Czechia
- France (2):
  - Centre Hospitalier Universitaire de Limoges, Department of Clinical Hematology and Cell Therapy, Limoges
  - Service de Néphrologie, Hémodialyse Et Transplantation Rénale, Hôpital Jean Bernard, Chu Poitiers, Poitiers
- Universität Heidelberg, Department of Internal Medicine V: Hematology, Oncology and Rheumatology, Heidelberg, Germany
- Alexandra Hospital, University of Athens School of Medicine, Department of Clinical Therapeutics, Athens, Greece
- Centro Per Lo Studio E La Cura Delle Amiloidosi Sistemiche Padiglione Forlanini, Pavia, Italy
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - University Medical Center Utrecht, Umc Utrecht, Department of Hematology, Utrecht
- Portugal (2):
  - Fundação Champalimaud, Hematology Research, Imunology - Medical School, Nova University, Lisbon
  - Centro Hospitalar E Universitário São João, Porto
- Servicio de Hematología, Hospital Clínic de Barcelona, Barcelona, Spain
- University College London Medical School, Uk Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided